CLINICAL TRIAL: NCT04512313
Title: A Single-blinded Multicenter Randomized Interventional Study of Rocuronium 0.3 mg/kg, and 0.9 mg/kg Comparing Onset Time, Duration of Action and Effect on Intubating Conditions in Elderly Patients (≥ 80 Years).
Brief Title: A Comparison of Rocuronium 0.3 mg/kg, and 0.9 mg/kg for Induction of Anesthesia in Elderly Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Matias Vested, Principal Investigator, Anesthesiologist, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-19079175
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Neuromuscular Blockade; Neuromuscular Blockade, Residual; Anesthesia; Intubation Complication
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving rocuronium 0,3 mg/kg (Active Comparator): Rocuronium 0,3 mg/kg at induction
  Interventions: Drug: Rocuronium 0,3mg/kg
- Group receiving rocuronium 0,9 mg/kg (Active Comparator): Rocuronium 0,9 mg/kg at induction
  Interventions: Drug: Rocuronium 0,9mg/kg

INTERVENTIONS:
Drug: Rocuronium 0,3mg/kg — Rocuronium 0,3mg/kg at induction
  Other Names: Rocuronium
  Arms: Group receiving rocuronium 0,3 mg/kg
Drug: Rocuronium 0,9mg/kg — Rocuronium 0,9mg/kg at induction
  Other Names: Rocuronium
  Arms: Group receiving rocuronium 0,9 mg/kg

SUMMARY:
The number of elderly patients above 80 years is increasing and a large proportion of these patients will require surgery and anesthesia.

During anesthesia neuromuscular blocking agents (NMBA) are administered to facilitate intubating conditions and reduce the trauma to the larynx and vocal cords. There is a risk of residual neuromuscular block when using NMBAs like rocuronium.

The aim of this study is to determine the onset time, duration of action and effect on intubating conditions after rocuronium 0.3 mg/kg and 0.9 mg/kg in patients with age ≥ 80 years.

DETAILED DESCRIPTION:
The number of elderly patients (>80 years) is increasing and a large proportion of these patients will require surgery and anesthesia within the next decades. Elderly patients are at higher risk of major morbidity and mortality and are characterized by a reduction in cardiac output, liver function and renal function. These physiological changes influence pharmacodynamics and pharmacokinetics of drugs administered during anesthesia.

Rocuronium is a nondepolarizing neuromuscular blocking drug with an onset time of approximately 70 s and a clinical duration of action of approximately 50 min. according to previous studies. During anesthesia rocuronium is administered to facilitate intubating conditions and reduce the trauma to the larynx and vocal cords. Rocuronium is primarily metabolized in the liver (70 % unmetabolized via the bile) and excreted via the kidneys.

Onset time and duration of action of rocuronium should be assessed by objective neuromuscular monitoring. Also, this reduces the risk of residual neuromuscular block which is defined as a train of four (TOF) ratio less than 0.9. Especially elderly patients have a high incidence of residual neuromuscular block.

The collected data regarding the effect of rocuronium in elderly patients may change the treatment so these patients receive the correct dose for optimal intubating conditions. Also, detection of duration of action of different doses of rocuronium may reduce the risk of residual block and postoperative respiratory complications

The aim of this study is to determine the onset time, duration of action and effect on intubating conditions after rocuronium 0.3 mg/kg and 0.9 mg/kg in patients with age ≥ 80 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80
* Scheduled to elective surgery (expected duration time of surgery > 1 hour) under general anesthesia with intubation and use of rocuronium.
* American Society of Anesthesiologists (ASA) physical status classification I to III
* Informed consent (see appendix 1)
* Read and understand Danish

Exclusion Criteria:

* Neuromuscular disease
* Known allergy to rocuronium
* Prone position
* Indication for rapid sequence induction

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Rocuronium onset time | intraoperative (From start of rocuronium injection to train-of-four (TOF) count of 0)
  Time from start of rocuronium injection to train-of-four (TOF) count of 0

SECONDARY OUTCOMES:
Duration of action of rocuronium | intraoperative (Time from start of rocuronium injection to reappearance of TOF ratio > 0.9.)
  Time from start of rocuronium injection to reappearance of TOF ratio > 0.9.
Evaluation of intubating conditions ad modum Fuchs-Buder et al | intraoperative (From train-of-four (TOF) count of 0 till)
  Intubating conditions are rated by an intubating difficulty scale according to Fuchs-Buder et al.

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, MD, PhD, Principal Investigator — Department of Anaesthesia, Head and Orthopaedics Centre, Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wadland SS, Rasmussen LS, Vested M. Shortened time to neuromuscular recovery with lower doses of rocuronium in elderly patients. Dan Med J. 2024 May 13;71(6):A09230578. doi: 10.61409/A09230578. PMID 38847412